CLINICAL TRIAL: NCT05979623
Title: Clinicopathological Characteristics and Prognosis Analysis of Stage IB Non-small Cell Lung Cancer：A Retrospective Real World Study
Brief Title: Clinicopathological Characteristics and Prognosis Analysis of Stage IB Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-128
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Stage IB Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ZS-IB-NSCLC: A total of 971 NSCLC patients with pathological stage IB resected by surgery (R0) from January 2016 to December 2020 at Zhongshan Hospital of Fudan University

SUMMARY:
The goal of this observation study is to learn about clinicopathological characteristics and prognostic factors of stage IB NSCLC. The main question it aims to answer is wheather there is relationship between newly proposed clinicopathological features and the prognosis of stage IB NSCLC .The postoperative pathological and follow-up information of participants will be used for subsequent analysis.

DETAILED DESCRIPTION:
A total of 971 NSCLC patients with pathological stage IB resected by surgery (R0) from January 2016 to December 2020 at Zhongshan Hospital of Fudan University were reviewed. The primary endpoint is RFS (recurrence-free survival) and OS (overall survival) is the secondary endpoint. The baseline characteristics of the patients were obtained statistically, and factors affecting the prognosis of patients with stage IB NSCLC were analyzed using survival analysis and Cox proportional hazard models. The characteristics of the patients include pathological type, STAS, GGO, gene mutation, and postoperative adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* It was confirmed by histopathology as primary non-small cell lung cancer, and the pathological type was LUSC or LUAD;
* According to the 8th edition of TNM clinical staging standards, it is determined as IB stage
* No treatment was performed for the primary lesion of lung cancer before surgery;
* No history of other malignant tumors before surgery;
* Detailed clinical and pathological information, complete survival data, and no missing follow-up data.

Exclusion Criteria:

* The postoperative histopathological types include non-scale and non adenocarcinoma, such as lung adenosquamous cell carcinoma, large cell lung cancer, or lung sarcomatoid carcinoma;
* Multiple lesion staging surgery;
* History of merging with other malignant tumors
* Having preoperative treatment;
* Missing follow-up information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients with pathological stage IB resected by surgery (R0)
Sampling Method: Non-Probability Sample
Enrollment: 971 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
RFS | 5 years
  recurrence-free survival

SECONDARY OUTCOMES:
OS | 5 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Di Ge, Ph.D;M.D, Study Chair — Zhongshan Hospital, Fudan University, Shanghai, China
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No